CLINICAL TRIAL: NCT03570047
Title: SAFETY AND EFFECTIVENESS EVALUATION OF PATIENTS WITH NON-VALVULAR ATRIAL FIBRILLATION TREATED WITH OACS: COMPARISON BETWEEN NOACS AND WARFARIN (CER3)
Brief Title: Safety and Effectiveness of Oral Anticoagulants in Patients With Non-valvular Atrial Fibrillation
Acronym: CER3
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B0661120; CER3 (Other: Alias Study Number)
Record Dates: First submitted 2018-06-15; First posted 2018-06-26 (Actual); Results first posted 2019-11-04 (Actual); Last update posted 2019-11-04 (Actual); Status verified 2019-10

CONDITIONS: Non-valvular Atrial Fibrillation
Keywords: Non-valvular atrial fibrillation, NVAF

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
An anticoagulation therapy is a critical treatment to prevent thromboembolism in non-valvular AF (NVAF) patients. Warfarin, a vitamin K antagonist, is the first oral anticoagulant approved for the treatment for prevention of thromboembolism and it had long been the only oral anticoagulant until the first non-vitamin K antagonist oral anticoagulants (NOACs). However, its safety and effectiveness remains unknown in real-world clinical practice in Japan

DETAILED DESCRIPTION:
An anticoagulation therapy is a critical treatment to prevent thromboembolism in non-valvular AF (NVAF) patients. Warfarin, a vitamin K antagonist, is the first oral anticoagulant approved for the treatment for prevention of thromboembolism and it had long been the only oral anticoagulant until the first non-vitamin K antagonist oral anticoagulants (NOACs). However, its safety and effectiveness remains unknown in real-world clinical practice in Japan. This study will evaluate the risk of stroke/SE as well as the risk of bleeding in the real world settings in Japan in patients with NVAF who initiated any of OACs (apixaban, dabigatran, edoxaban, rivaroxaban, or warfarin)

ELIGIBILITY:
Inclusion criteria

Patients must meet all of the following criteria to be eligible for the study:

1. Diagnosed with AF anytime in the baseline period or on the index date, also have definitive diagnosis of AF anytime in the baseline period, on the index date, or post-index period.
2. Prescribed one of the index OACs (apixaban, dabigatran, edoxaban, rivaroxaban or warfarin) on or after the day of AF diagnosis. The first observed prescription will be used to identify the patient's index date and treatment cohort
3. No use of the any OACs during the baseline period (the 180 days before the index date)
4. Age of 18 years or older on the index date.

Exclusion criteria

Patients meeting any of the following criteria will not be included in the study:

1. Having a diagnosis of valvular atrial fibrillation, post-operative atrial fibrillation, rheumatic atrial fibrillation or mechanical-valvular atrial fibrillation during the baseline and post-index period 2. Having a cardiac surgery procedure record during the baseline period 3. Having a joint replacement procedure record during the baseline period 4. Having a procedure of prosthetic heart valve during the baseline period 5. Having a diagnosis of venous thromboembolism during the baseline period 6. Female patients with pregnancy during the follow-up period 7. Patients prescribed "off-label" doses of OACs (per Japanese package insert of each OAC) or patients treated with OAC but in "off-label" or "contraindicated" manners.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with NVAF who initiated any of oral anti-coagulants
Sampling Method: Non-Probability Sample
Enrollment: 73989 (Actual)
Dates: Start 2018-05-08 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Japan, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B0661120

RESULTS

PARTICIPANT FLOW:
Recruitment Details: It is a retrospective population-based register study. Data of each participant diagnosed with non-valvular atrial fibrillation (NAVF) was retrieved from Medical Data Vision (MDV) database for the duration of approximately 7 years (March 2011 to December 2017).
Pre-assignment Details: In this study, inverse probability of treatment weighted (IPTW) method was used in analysis of outcome measures to balance participant's characteristics among reporting groups.
Groups:
- Warfarin: Oral anticoagulants (OACs) treatment-naive participants diagnosed with NVAF, who initiated warfarin on the index date, were included in this study cohort and their data (for the duration of approximately 7 years observation period, i.e. 2011-2017) available in MDV database was retrospectively observed. Index date was defined as the date of the first prescription of any OACs (warfarin, apixaban, dabigatran, rivaroxaban or edoxaban) during observation period.
- Apixaban: OACs treatment-naive participants diagnosed with NVAF, who initiated apixaban on the index date, were included in this study cohort and their data (for the duration of approximately 7 years observation period, i.e. 2011-2017) available in MDV database was retrospectively observed. Index date was defined as the date of the first prescription of any OACs (warfarin, apixaban, dabigatran, rivaroxaban or edoxaban) during observation period.
- Dabigatran: OACs treatment-naive participants diagnosed with NVAF, who initiated dabigatran on the index date, were included in this study cohort and their data (for the duration of approximately 7 years observation period, i.e. 2011-2017) available in MDV database was retrospectively observed. Index date was defined as the date of the first prescription of any OACs (warfarin, apixaban, dabigatran, rivaroxaban or edoxaban) during observation period.
- Rivaroxaban: OACs treatment-naive participants diagnosed with NVAF, who initiated rivaroxaban on the index date, were included in this study cohort and their data (for the duration of approximately 7 years observation period, i.e. 2011-2017) available in MDV database was retrospectively observed. Index date was defined as the date of the first prescription of any OACs (warfarin, apixaban, dabigatran, rivaroxaban or edoxaban) during observation period.
- Edoxaban: OACs treatment-naive participants diagnosed with NVAF, who initiated edoxaban on the index date, were included in this study cohort and their data (for the duration of approximately 7 years observation period, i.e. 2011-2017) available in MDV database was retrospectively observed. Index date was defined as the date of the first prescription of any OACs (warfarin, apixaban, dabigatran, rivaroxaban or edoxaban) during observation period.
Period: Overall Study
Arm/Group | Warfarin | Apixaban | Dabigatran | Rivaroxaban | Edoxaban
Started | 15902 | 22336 | 6925 | 16564 | 12262
Completed | 15902 | 22336 | 6925 | 16564 | 12262
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: OACs treatment-naive participants diagnosed with NVAF initiating any OACs (warfarin, apixaban, dabigatran, rivaroxaban or edoxaban) treatment were included in the study.
Groups:
- Warfarin: OACs treatment-naive participants diagnosed with NVAF, who initiated warfarin on the index date, were included in this study cohort and their data (for the duration of approximately 7 years observation period, i.e. 2011-2017) available in MDV database was retrospectively observed. Index date was defined as the date of the first prescription of any OACs (warfarin, apixaban, dabigatran, rivaroxaban or edoxaban) during observation period.
- Total: Total of all reporting groups
Arm/Group | Warfarin | Apixaban | Dabigatran | Rivaroxaban | Edoxaban | Total
Number analyzed (Participants) | 15902 | 22336 | 6925 | 16564 | 12262 | 73989
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1312 | 2298 | 1331 | 2705 | 1451 | 9097
  >=65 years | 14590 | 20038 | 5594 | 13859 | 10811 | 64892
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6257 | 9131 | 2184 | 5818 | 5331 | 28721
  Male | 9645 | 13205 | 4741 | 10746 | 6931 | 45268
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Event Rate Per 100 Participant-Years For First Occurrence of Stroke and Systemic Embolism Events After Index Date
Description: Event rate per 100 participant-years for first occurrence of stroke and systemic embolism events after index date was reported. Stroke events included the composite of any ischemic and any hemorrhagic stroke events (non-traumatic extradural hemorrhage). Systemic embolism events were defined as any of the following: abdominal aortic embolism, aortic embolism, acute arterial occlusive disease of arteries of upper extremities, femoral arterial occlusion and acute arterial occlusive disease of arteries of lower extremities, iliac artery embolism, hepatic artery embolism, thromboembolism, embolic infarction, aortic embolism, subclavian artery stenosis. Index date was defined as date of first prescription of any OACs (warfarin, apixaban, dabigatran, rivaroxaban or edoxaban) during the observation period of approximately 7 years (2011-2017). Pseudo datasets refers to number derived using IPTW method and are different from the actual participants included in the reporting arm.
Time Frame: During the observation period of approximately 7 years
Population: OACs treatment-naive participants diagnosed with NVAF, initiating any OACs treatment were included in study. Analysis performed using IPTW method to balance participant characteristics among reporting groups. IPTW method created weighted pseudo-datasets which were used in analysis of outcome measure and are reported in the "units analyzed" field.
Measure: Number; unit: Events Per 100 Participant-Years
Units Other Than Participants: Pseudo datasets
Arm/Group | Warfarin | Apixaban | Dabigatran | Rivaroxaban | Edoxaban
Number analyzed (Participants) | 15902 | 22336 | 6925 | 16564 | 12262
Number analyzed (Pseudo datasets) | 19059 | 22752 | 8003 | 17481 | 12592
Events Per 100 Participant-Years | 3.2 | 1.67 | 2.08 | 1.79 | 2
Statistical Analysis 1: Comparison: Warfarin vs Apixaban; Test type: Other; p < 0.0001, Cox proportional hazards model; Hazard Ratio (HR) = 0.65, 95% CI 2-sided [0.558 to 0.766]
Statistical Analysis 2: Comparison: Warfarin vs Dabigatran; Test type: Other; p = 0.0291, Cox proportional hazards model; Hazard Ratio (HR) = 0.79, 95% CI 2-sided [0.642 to 0.977]
Statistical Analysis 3: Comparison: Warfarin vs Rivaroxaban; Test type: Other; p = 0.0001, Cox proportional hazards model; Hazard Ratio (HR) = 0.71, 95% CI 2-sided [0.592 to 0.842]
Statistical Analysis 4: Comparison: Warfarin vs Edoxaban; Test type: Other; p = 0.0012, Cox proportional hazards model; Hazard Ratio (HR) = 0.72, 95% CI 2-sided [0.591 to 0.879]

2. Primary Outcome: Event Rate Per 100 Participant-Years For First Occurrence of Major Bleeding Events After Index Date
Description: Event rate per 100 participant-years for first occurrence of major bleeding event after index date was reported. Major bleeding after index date was identified using hospital claims which had a bleeding diagnosis code as the first listed in International Statistical Classification of Diseases and Related Health Problems (ICD)-10 diagnosis code. An event occurrence of major bleeding was defined as that appears as "21: Disease name behind hospitalization" in database. Index date was defined as the date of the first prescription of any of OACs (warfarin, apixaban, dabigatran, rivaroxaban or edoxaban) during the observation period of approximately 7 years (2011-2017). Pseudo datasets refers to number derived using IPTW method and are different from the actual participants included in the reporting arm.
Time Frame: During the observation period of approximately 7 years
Population: as for outcome 1
Measure: Number; unit: Events Per 100 Participant-Years
Units Other Than Participants: Pseudo datasets
Arm/Group | Warfarin | Apixaban | Dabigatran | Rivaroxaban | Edoxaban
Number analyzed (Participants) | 15902 | 22336 | 6925 | 16564 | 12262
Number analyzed (Pseudo datasets) | 19059 | 22752 | 8003 | 17481 | 12592
Events Per 100 Participant-Years | 3.13 | 1.79 | 1.72 | 1.82 | 1.91
Statistical Analysis 1: Comparison: Warfarin vs Apixaban; Test type: Other; p < 0.0001, Cox proportional hazards model; Hazard Ratio (HR) = 0.72, 95% CI 2-sided [0.614 to 0.843]
Statistical Analysis 2: Comparison: Warfarin vs Dabigatran; Test type: Other; p = 0.0003, Cox proportional hazards model; Hazard Ratio (HR) = 0.66, 95% CI 2-sided [0.529 to 0.825]
Statistical Analysis 3: Comparison: Warfarin vs Rivaroxaban; Test type: Other; p = 0.0007, Cox proportional hazards model; Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.618 to 0.879]
Statistical Analysis 4: Comparison: Warfarin vs Edoxaban; Test type: Other; p = 0.0011, Cox proportional hazards model; Hazard Ratio (HR) = 0.71, 95% CI 2-sided [0.583 to 0.874]

3. Primary Outcome: Event Rate Per 100 Participant-Years For First Occurrence of Any Bleeding Event After Index Date
Description: Event rate per 100 participant-years for first occurrence of any bleeding event after index date was reported. Any bleeding was defined using ICD-10 diagnosis codes and participants were considered to have "any bleeding" if pre-defined bleeding-associated ICD-10 diagnosis codes appeared in the records. Index date was defined as the date of the first prescription of any of OACs (warfarin, apixaban, dabigatran, rivaroxaban or edoxaban) during the observation period of approximately 7 years (2011-2017). Pseudo datasets refers to number derived using IPTW method and are different from the actual participants included in the reporting arm.
Time Frame: During the observation period of approximately 7 years
Population: as for outcome 1
Measure: Number; unit: Events Per 100 Participant-Years
Units Other Than Participants: Pseudo datasets
Arm/Group | Warfarin | Apixaban | Dabigatran | Rivaroxaban | Edoxaban
Number analyzed (Participants) | 15902 | 22336 | 6925 | 16564 | 12262
Number analyzed (Pseudo datasets) | 19059 | 22752 | 8003 | 17481 | 12592
Events Per 100 Participant-Years | 22.11 | 15.97 | 15.9 | 16.07 | 20.34
Statistical Analysis 1: Comparison: Warfarin vs Apixaban; Test type: Other; p = 0.0127, Cox proportional hazards model; Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.872 to 0.984]
Statistical Analysis 2: Comparison: Warfarin vs Dabigatran; Test type: Other; p = 0.2893, Cox proportional hazards model; Hazard Ratio (HR) = 0.96, 95% CI [0.881 to 1.039]
Statistical Analysis 3: Comparison: Warfarin vs Rivaroxaban; Test type: Other; p = 0.0640, Cox proportional hazards model; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.881 to 1.004]
Statistical Analysis 4: Comparison: Warfarin vs Edoxaban; Test type: Other; p = 0.4404, Cox proportional hazards model; Hazard Ratio (HR) = 1.03, 95% CI 2-sided [0.958 to 1.103]

4. Secondary Outcome: Event Rate Per 100 Participant-Years For First Occurrence of Ischemic Stroke After Index Date
Description: Event rate per 100 participant-years for first occurrence of ischemic stroke after index date was reported. Index date was defined as the date of the first prescription of any of OACs (warfarin, apixaban, dabigatran, rivaroxaban or edoxaban) during the observation period of approximately 7 years (2011-2017). Pseudo datasets refers to number derived using IPTW method and are different from the actual participants included in the reporting arm.
Time Frame: During the observation period of approximately 7 years
Population: as for outcome 1
Measure: Number; unit: Events Per 100 Participant-Years
Units Other Than Participants: Pseudo datasets
Arm/Group | Warfarin | Apixaban | Dabigatran | Rivaroxaban | Edoxaban
Number analyzed (Participants) | 15902 | 22336 | 6925 | 16564 | 12262
Number analyzed (Pseudo datasets) | 19059 | 22752 | 8003 | 17481 | 12592
Events Per 100 Participant-Years | 2.4 | 1.2 | 1.76 | 1.41 | 1.54

5. Secondary Outcome: Event Rate Per 100 Participant-Years For First Occurrence of Hemorrhagic Stroke After Index Date
Description: Event rate per 100 participant-years for first occurrence of hemorrhagic stroke after index date was reported. Index date was defined as the date of the first prescription of any of OACs (warfarin, apixaban, dabigatran, rivaroxaban or edoxaban) during the observation period of approximately 7 years (2011-2017). Pseudo datasets refers to number derived using IPTW method and are different from the actual participants included in the reporting arm.
Time Frame: During the observation period of approximately 7 years
Population: as for outcome 1
Measure: Number; unit: Events Per 100 Participant-Years
Units Other Than Participants: Pseudo datasets
Arm/Group | Warfarin | Apixaban | Dabigatran | Rivaroxaban | Edoxaban
Number analyzed (Participants) | 15902 | 22336 | 6925 | 16564 | 12262
Number analyzed (Pseudo datasets) | 19059 | 22752 | 8003 | 17481 | 12592
Events Per 100 Participant-Years | 0.72 | 0.43 | 0.25 | 0.36 | 0.43

6. Secondary Outcome: Event Rate Per 100 Participant-Years For First Occurrence of Systemic Embolism Events After Index Date
Description: Event rate per 100 participant-years for first occurrence of systemic embolism events after index date was reported. Systemic embolism events included any of the following: abdominal aortic embolism, aortic embolism, acute arterial occlusive disease of arteries of upper extremities, femoral arterial occlusion and acute arterial occlusive disease of arteries of lower extremities, iliac artery embolism, hepatic artery embolism, thromboembolism, embolic infarction, aortic embolism, subclavian artery stenosis. Index date was defined as the date of the first prescription of any of OACs (warfarin, apixaban, dabigatran, rivaroxaban or edoxaban) during the observation period of approximately 7 years (2011-2017). Pseudo datasets refers to number derived using IPTW method and are different from the actual participants included in the reporting arm.
Time Frame: During the observation period of approximately 7 years
Population: as for outcome 1
Measure: Number; unit: Events Per 100 Participant-Years
Units Other Than Participants: Pseudo datasets
Arm/Group | Warfarin | Apixaban | Dabigatran | Rivaroxaban | Edoxaban
Number analyzed (Participants) | 15902 | 22336 | 6925 | 16564 | 12262
Number analyzed (Pseudo datasets) | 19059 | 22752 | 8003 | 17481 | 12592
Events Per 100 Participant-Years | 0.11 | 0.04 | 0.08 | 0.04 | 0.05

7. Secondary Outcome: Event Rate Per 100 Participant-Years For First Occurrence of Major Gastrointestinal Bleeding Events After Index Date
Description: Event rate per 100 participant-years for first occurrence of major gastrointestinal bleeding events after index date was reported. Major gastrointestinal bleeding after index date was identified using hospital claims which had a gastrointestinal bleeding diagnosis code as the first listed ICD-10 diagnosis code. An event occurrence of major bleeding was defined as that appears as "21: Disease name behind hospitalization" in database. Index date was defined as the date of the first prescription of any of OACs (warfarin, apixaban, dabigatran, rivaroxaban or edoxaban) during the observation period of approximately 7 years (2011-2017). Pseudo datasets refers to number derived using IPTW method and are different from the actual participants included in the reporting arm.
Time Frame: During the observation period of approximately 7 years
Population: as for outcome 1
Measure: Number; unit: Events Per 100 Participant-Years
Units Other Than Participants: Pseudo datasets
Arm/Group | Warfarin | Apixaban | Dabigatran | Rivaroxaban | Edoxaban
Number analyzed (Participants) | 15902 | 22336 | 6925 | 16564 | 12262
Number analyzed (Pseudo datasets) | 19059 | 22752 | 8003 | 17481 | 12592
Events Per 100 Participant-Years | 1.02 | 0.61 | 0.77 | 0.74 | 0.73

8. Secondary Outcome: Event Rate Per 100 Participant-Years For First Occurrence of Any Gastrointestinal Bleeding Event After Index Date
Description: Event rate per 100 participant-years for first occurrence of any gastrointestinal bleeding event after index date was reported. Any gastrointestinal bleeding was defined by ICD-10 diagnosis codes. If participants had ICD-10 diagnosis codes which suggest bleeding from the gastrointestinal tract, they were considered to have any gastrointestinal bleeding. Index date was defined as the date of the first prescription of any of OACs (warfarin, apixaban, dabigatran, rivaroxaban or edoxaban) during the observation period of approximately 7 years (2011-2017). Pseudo datasets refers to number derived using IPTW method and are different from the actual participants included in the reporting arm.
Time Frame: During the observation period of approximately 7 years
Population: as for outcome 1
Measure: Number; unit: Events Per 100 Participant-Years
Units Other Than Participants: Pseudo datasets
Arm/Group | Warfarin | Apixaban | Dabigatran | Rivaroxaban | Edoxaban
Number analyzed (Participants) | 15902 | 22336 | 6925 | 16564 | 12262
Number analyzed (Pseudo datasets) | 19059 | 22752 | 8003 | 17481 | 12592
Events Per 100 Participant-Years | 5.98 | 4.11 | 4.75 | 4.07 | 5.42

9. Secondary Outcome: Event Rate Per 100 Participant-Years For First Occurrence of Major Intracranial Hemorrhage Events After Index Date
Description: Event rate per 100 participant-years for first occurrence of major intracranial hemorrhage events after index date was reported. Major intracranial hemorrhage was defined by ICD-10 diagnosis codes and participants were considered to have "major intracranial hemorrhage" if pre-defined major intracranial hemorrhagic-associated ICD-10 diagnosis codes appeared in the records. Index date was defined as the date of the first prescription of any of OACs (warfarin, apixaban, dabigatran, rivaroxaban or edoxaban) during the observation period of approximately 7 years (2011-2017). Pseudo datasets refers to number derived using IPTW method and are different from the actual participants included in the reporting arm.
Time Frame: During the observation period of approximately 7 years
Population: as for outcome 1
Measure: Number; unit: Events Per 100 Participant-Years
Units Other Than Participants: Pseudo datasets
Arm/Group | Warfarin | Apixaban | Dabigatran | Rivaroxaban | Edoxaban
Number analyzed (Participants) | 15902 | 22336 | 6925 | 16564 | 12262
Number analyzed (Pseudo datasets) | 19059 | 22752 | 8003 | 17481 | 12592
Events Per 100 Participant-Years | 1.22 | 0.57 | 0.43 | 0.5 | 0.62

10. Secondary Outcome: Event Rate Per 100 Participant-Years For First Occurrence of Any Intracranial Hemorrhage Event After Index Date
Description: Event rate per 100 participant-years for first occurrence of any intracranial hemorrhage event after index date was reported. Any intracranial hemorrhage was defined by ICD-10 diagnosis codes and participants were considered to have "any intracranial hemorrhagic event" if pre-defined any intracranial hemorrhagic-associated ICD-10 diagnosis codes appeared in the records. Index date was defined as the date of the first prescription of any of OACs (warfarin, apixaban, dabigatran, rivaroxaban or edoxaban) during the observation period of approximately 7 years (2011-2017). Pseudo datasets refers to number derived using IPTW method and are different from the actual participants included in the reporting arm.
Time Frame: During the observation period of approximately 7 years
Population: as for outcome 1
Measure: Number; unit: Events Per 100 Participant-Years
Units Other Than Participants: Pseudo datasets
Arm/Group | Warfarin | Apixaban | Dabigatran | Rivaroxaban | Edoxaban
Number analyzed (Participants) | 15902 | 22336 | 6925 | 16564 | 12262
Number analyzed (Pseudo datasets) | 19059 | 22752 | 8003 | 17481 | 12592
Events Per 100 Participant-Years | 4.16 | 2.93 | 2.43 | 2.66 | 3.65

ADVERSE EVENTS:
Description: Due to observational nature of study, adverse events were not collected in this study.
Arm/Group | Warfarin | Apixaban | Dabigatran | Rivaroxaban | Edoxaban
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2018-05-08): https://cdn.clinicaltrials.gov/large-docs/47/NCT03570047/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-14): https://cdn.clinicaltrials.gov/large-docs/47/NCT03570047/SAP_001.pdf